CLINICAL TRIAL: NCT00329862
Title: Pilot Study Assessing Advantage of Adding Truncal Vagotomy to LAGB
Brief Title: Laparoscopic Adjustable Gastric Banding With Truncal Vagotomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study size reached
Sponsor: Central Carolina Surgery, PA (Other)
Collaborators: EndoVx, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAGBTV
Record Dates: First submitted 2006-05-23; First posted 2006-05-25 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: Morbid Obesity; Obstructive Sleep Apnea; Hypertension; Urinary Incontinence; Hypertriglyceridemia; Diabetes; Hypercholesterolemia
Keywords: Laparoscopic Adjustable Gastric Banding; Truncal Vagotomy; Lap Band; Lap Banding; Obesity Surgery; Bariatric surgery; Weight Loss Surgery
MeSH Terms: conditions — Obesity, Morbid; Sleep Apnea, Obstructive; Hypertension; Urinary Incontinence; Hypertriglyceridemia; Diabetes Mellitus; Hypercholesterolemia

INTERVENTIONS:
Procedure: Laparoscopic Truncal Vagotomy

SUMMARY:
Laparoscopic Adjustable Gastric Banding (LAGB) is a gold standard in the surgical treatment of morbid obesity. We hypothesize that the addition of truncal vagotomy (cutting of nerves to the stomach) will produce greater weight loss and better reduction of co-morbidities (diseases caused by or aggravated by morbid obesity) than LAGB alone. 25 patients will be enrolled and outcomes compared to LAGB historical controls over a post-operative period of 24 months.

DETAILED DESCRIPTION:
The patients will receive standard laparoscopic adjustable gastric banding treatment as well as truncal vagotomy. The vagus nerves will be cut just below the diaphragm using the same access ports that are used during the laparoscopic adjustable gastric banding. During the surgical procedure, the first fifteen patients will also receive a dose of Baclofen, a vagus nerve stimulant, and an endoscopy at the end of the procedure during which congo red dye will sprayed within the stomach. The Baclofen and endoscopy are used to ensure that all branches of the vagus nerve have been cut. If, after 15 complete vagotomies, are verified by the above testing then the use of Baclofen and endoscopy will be abandoned.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient between 18 to 60 years of age.
2. Patient has body mass index (BMI) between 40 to 50 or a BMI between 35 to 40 with one or more co-morbidities , and a stable weight for the last 3 months (+ 3 kg).
3. Female patients must be willing to use contraceptive methods during the course of the trial (18 months).
4. Patient must be motivated to lose weight.
5. Patient has a history of at least one professionally supervised 6 month attempt to lose weight or more than two serious attempts.
6. Patient must be fully ambulatory.
7. Patient is to sign and be given a copy of the written informed consent form. -

Exclusion Criteria:

1. History or signs of prior gastric or esophageal surgery
2. History of or signs and/or symptoms of gastro-duodenal ulcer disease.
3. Participation or plans for participation in another investigational study during the study period.
4. Patients with large hiatal hernias. -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-05; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Excess body weight loss measured @ 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 weeks
BMI reduction measured @ 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 weeks
Reduction and or elimination of co-morbidities @ 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Hardcastle, MD, Principal Investigator — Central Carolina Surgery, PA